CLINICAL TRIAL: NCT01880931
Title: The Effect Site Concentration of Remifentanil for Preventing QTc Interval Prolongation During Intubation in Normotensive and Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2013-0239
Record Dates: First submitted 2013-06-16; First posted 2013-06-19 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Intubation, Intratracheal
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normotensive patients (Experimental): To find out the effect site concentration of remifentanil for preventing QTc prolongation < 15 sec during intubation : Dixon's up-and-down method
  Interventions: Drug: Remifentanil
- Hypertensive patients (Experimental): To find out the effect site concentration of remifentanil for preventing QTc prolongation < 15 sec during intubation : Dixon's up-and-down method
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — The effect site concentration of remifentanil

SUMMARY:
To find out the effect site concentration of remifentanil for preventing QTc interval prolongation during intubation under propofol-remifentanil anesthesia in normotensive and hypertensive patients

DETAILED DESCRIPTION:
It is known that anesthetic agents can influence the QTc. In addition, tracheal intubation during induction can stimulates sympathetic activity, which, as a results, prolong the QTc interval. Therefore, the aim of study is to find out the effect site concentration of remifentanil for preventing QTc interval prolongation during intubation under propofol-remifentanil anesthesia in normotensive and hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years ASA class I-II female who received surgery with endotracheal intubation

Exclusion Criteria:

* emergency surgery electrocardiography abnormality diabetes mellitus end stage renal disease moderate to severe cardiac disease moderate to severe liver dysfunction

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
The effect site concentration of remifentanil for preventing QTc interval prolongation | 2 min

CONTACTS AND LOCATIONS:
Overall Officials: So Yeon Kim, MD, PhD, Principal Investigator — Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea